CLINICAL TRIAL: NCT00095771
Title: A Phase I Trial of Arsenic Trioxide in the Treatment of Infiltrating Gliomas of Childhood
Brief Title: Arsenic Trioxide and Radiation Therapy in Treating Young Patients With Newly Diagnosed Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000393829; P30CA006973 (NIH); JHOC-J0423; JHOC-04041906
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma; childhood high-grade cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Arsenic Trioxide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells and may be an effective treatment for patients with glioma. Drugs such as arsenic trioxide may also make the tumor cells more sensitive to radiation therapy. Combining arsenic trioxide with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining arsenic trioxide with radiation therapy in treating patients who have newly diagnosed gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of arsenic trioxide when administered with radiotherapy in pediatric patients with newly diagnosed anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, or intrinsic pontine glioma.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of arsenic trioxide (ATO).

Patients undergo radiotherapy once daily, 5 days a week, for approximately 6 weeks. Patients concurrently receive ATO IV over 1 hour, 1-5 times weekly, for approximately 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ATO until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 3-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Clinical and neuroradiographic findings consistent with intrinsic pontine glioma
  * Histologically confirmed anaplastic astrocytoma, glioblastoma multiforme, or gliosarcoma

    * Multifocal high-grade gliomas allowed
* No exophytic tumors
* No focal lesions
* No underlying diagnosis of neurofibromatosis
* No tumors originating in anatomic structures adjacent to the cerebellar peduncle or cervical medullary junction

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Karnofsky 60-100% OR
* Lansky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin > 10 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 2.0 mg/dL
* Alkaline phosphatase < 2.5 times upper limit of normal (ULN)
* Transaminases < 2.5 times ULN

Renal

* Creatinine < 2.0 times ULN

Cardiovascular

* No second-degree heart block
* No absolute QTc interval > 500 msec with normal potassium and magnesium levels

Other

* Not pregnant or nursing
* Negative pregnancy test
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ
* No other serious medical illness
* Able to undergo MRI

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* No prior arsenic trioxide

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Prior surgery for the brain tumor allowed

Other

* No other prior therapy for the brain tumor
* More than 28 days since prior investigational drugs or devices
* No concurrent amphotericin B

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose as assessed by NCI CTCAE v. 3.0 following study completion
Safety as assessed by NCI CTCAE v. 3.0 following study completion

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Cohen, MD, MBA, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States